CLINICAL TRIAL: NCT04392128
Title: Randomised, Double-blind, Placebo-controlled Phase 2 Study Evaluating the Efficacy of Hydroxychloroquine and Azithromycine in Patients With COVID-19 and Hematological Malignancies
Brief Title: Study Evaluating the Efficacy of Hydroxychloroquine and Azithromycine in Patients With COVID-19 and Hematological Malignancies (HYACINTHE)
Acronym: HYACINTHE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: competent authority decision
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-005; 2020-002002-45 (EudraCT Number)
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: COVID19; Hematologic Malignancy
Keywords: SARS-CoV-2; Hematologic malignancy
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Patients enrolled in the experimental arm will receive hydroxychloroquine (200mgx3 tablets per day during 10 days) and azithromycine (500 mg at day 1 (2 capsules taken at the same time) then 250mg per day (1 capsule per day) during 4 days).
  Interventions: Drug: Hydroxychloroquine Sulfate 200 MG [Plaquenil]; Drug: Azithromycin 250 MG Oral Capsule
- Control arm (Placebo Comparator): Patients enrolled in the control arm will receive a placebo of hydroxychloroquine (3 tablets per day during 10 days) and a placebo of azithromycine (2 capsules taken at the same time at day 1, then 1 capsule per day during 4 days)
  Interventions: Drug: Placebo oral tablet; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 200 MG [Plaquenil] — Hydroxychloroquine is an anti-malarial drug also used as anti-inflammatory treatment for systemic lupus erythematosus and rheumatic disorders. HCQ also inhibits pH-dependant replication stages of diverse types of viruses including flavivirus, retrovirus and coronaviruses.
  Arms: Treatment arm
Drug: Azithromycin 250 MG Oral Capsule — Azithromycin is amacrolide antibiotic.
  Arms: Treatment arm
Drug: Placebo oral tablet — Placebo of Hydroxychloroquine Sulfate 200 MG [Plaquenil].
  Arms: Control arm
Drug: Placebo oral capsule — Placebo of Azithromycin capsules.
  Arms: Control arm

SUMMARY:
The primary objective of this phase 2, multicentric, placebo-controlled double-blind, randomized study is to evaluate the efficacy of the combination of hydroxychloroquine and azithromycine on the viral load drop at day 5 among patients with COVID-19 and hematological malignancies.

DETAILED DESCRIPTION:
The study will evaluate the effect of the combination of hydroxychloroquine and azithromycine versus placebo among 114 patients with COVID-19 and hematologic malignancy.

After randomization in 1:1 ratio, patients will receive either the study treatment or placebo :

* Patients enrolled in the experimental arm will receive hydroxychloroquine (200mgx3 tablets per day during 10 days) and azithromycine (500 mg at day 1 then 250mg per day during 4 days)
* Patients enrolled in the control arm will receive a placebo of hydroxychloroquine (3 tablets per day during 10 days) and a placebo of azithromycine (2 capsules at day 1, then 1 capsule per day during 4 days)

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older patients
* Patient with hematologic malignancy who received or not hematopoietic stem cell transplantation
* Non severe Covid-19 disease
* PCR-confirmed COVID-19 disease by a nasopharyngeal swab
* Life-expectancy related to the hematologic malignancy of at least 1 month
* Men or women of child-bearing potential accepting to use effective contraception during and until 8 months after the end of the study treatment

Exclusion Criteria:

* Patients with severe form of COVID-19 infection defined as the presence of crackles observed during clinical exam, associated with less than 94% oxygen saturation or patients with respiratory insufficiency on oxygen therapy or mechanical ventilation
* Previous treatment with hydroxychloroquine or azithromycine for Covid-19 infection
* QTc interval greater than 480 ms
* Hypersensibility to hydroxychloroquine or azithromycine
* Retinopathy
* TGO or TGP geater than 5 x the normal upper limit
* Creatinine clearance lower than 30 ml/min
* Concomitant treatment that may lead to prolongation of the QT space
* Concomitant treatment with dihydroergotamine, ergotamine, cisapride or colchicine
* Known G6PD deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of hydroxychloroquine and azithromyncine on the viral load drop at day 5. | 5 days of treatment
  Locally evaluated rate of viral response. Favorable response is defined as (1) complete response : negative PCR (absence of detectable signal with a minimum of 40 cycles) or (2) major response : detectable signal but with an increased number of cycles > or egal to 10 compared to initial PCR. Response failure is defined as (1) minor response : detectable signal but with an increased number of cycles < 10 compared to initial PCR or (2) stabilisation or worsening of the viral load.

SECONDARY OUTCOMES:
Clinical evolution | up to 3 months
  Duration of fever - duration of respiratory symptoms (cough, dyspnea) - duration of other COVID-19 related symptoms (digestive symptoms, ageusia, anosmia)
Proportion of patients progressing to a severe form | up to 3 months
  Less or equal to 94% oxygen saturation - need to initiate oxygenotherapy - occurrence of respiratory distress - patient transfer in intensive care unit - need of mechanical ventilation - occurrence of non-respiratory organ failure - occurrence of septic shock
Mortality | up to 1 and 3 months
  Date and cause of death
Evaluation of viral load drop | at day 10
  SARS-CoV-2 viral load by PCR on nasopharyngeal swab at day 10 (if positive at day 5) : rate of negativation and comparison of number of cycles with previous samples
Tolerance of study treatment | up to 3 months
  Frequence and causality of all-grade cardiac adverse events - frequence and causality of grade > 1 adverse events for other adverse events - frequence and causality of serious adverse events (CTCAE v5)
Evaluation of the seroconversion | at inclusion, day 10, day 30 and day 90 after treatment
  Collection of serum to realize serological tests
NK immunological study | at day 10 and day 30 after treatment
  Phenotypic and functional study of NK lymphocytes at inclusion, Retrospective analysis on frozen cells.
Hospitalisation duration | up to 3 months
  Duration of hospitalisation (conventional, intensive care, reanimation)
Impact of the study treatment on the treatment of the hematological disease | up to 3 months
  Patient follow-up during 3 months : hematological status and associated therapy
Monitoring of the QT space | at inclusion, day 2, day 5, day 10
  ECG (using connected machine to allow monitoring at home)
Dosage of residual concentration of azithromycine and hydroxychloroquine. | at day 5 and day 10
  Dosage of residual concentration of azithromycine and hydroxychloroquine.
T immunological study | at day 10 and day 30 after treatment
  Phenotypic and functional study of T lymphocytes at inclusion, Retrospective analysis on frozen cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancérologie Strasbourg Europe, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No